CLINICAL TRIAL: NCT03132987
Title: Characterizing Clinical and Biomechanical Contributions to Function Following ACL Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Creighton University (Other)
Collaborators: University of Nebraska (Other); National Institutes of Health (NIH) (NIH); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 928791; 5P20GM109090-03 (NIH)
Record Dates: First submitted 2017-01-30; First posted 2017-04-28 (Actual); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: ACL Tears
Keywords: quadriceps strength; quadriceps voluntary activation; progressive strength program
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: Physical therapy exercises (progressive strengthening program)
Oversight: Data Monitoring Committee: No

ARMS (1):
- Progressive strengthening program (Experimental): Subjects identified as having a clinically relevant strength deficit will be asked to participate in physical therapy sessions 3 times per week for 3 weeks. The strengthening program will consist of an individualized, progressive exercise program with an emphasis on increasing lower extremity strength, power, and biomechanics.
  Interventions: Other: Progressive strengthening program

INTERVENTIONS:
Other: Progressive strengthening program — The progressive strengthening program will be performed for 3 weeks and emphasize development of strength and power. Feasibility will be established if we can recruit up to 8 participants and retain at least 80% over the 3 week intervention program. We will determine effect sizes for changes outcome measures.

SUMMARY:
Quantify differences in quadriceps function and gait biomechanics in individuals within 2 years of ACL reconstruction compared to a healthy comparison group and establish the feasibility of conducting a progressive strengthening program to improve clinical and patient-oriented outcomes in individuals who are within 2 years of ACL reconstruction

DETAILED DESCRIPTION:
A maximal isometric muscle contraction of the quadriceps will be used to examine neural and peripheral contributions to quadriceps strength. Neural influences will be quantified using the interpolated twitch technique (voluntary activation) and early RTD. Peripheral influences will be quantified by examining the stimulus-evoked torque with the quadriceps relaxed (resting twitch) and late RTD. Knee joint biomechanics during treadmill walking and running will include sagittal plane (flexion, extension) movement variability (Lyapunov Exponent and approximate entropy), peak knee flexion angle, and peak external knee flexion and adduction moments. Additionally, the clinical relevance of impairments in the ACL reconstruction group will be determined by examining the relationship with performance on jumping tasks and patient function (secondary outcomes).

The progressive strengthening program will be performed for 6 weeks and emphasize development of strength and power. Feasibility will be established if the researchers can recruit up to 8 participants and retain at least 80% over the 3 week intervention program. The researchers will determine effect sizes for changes outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Physically active
* History of primary unilateral ACL reconstruction within the past 3-24 months (ACL group only)

Exclusion Criteria:

* History of lumbar spine or lower extremity injury or surgery (except ACL) within the past 1 year that required physician care
* Concomitant knee injury (ACL group only): ligament injury that requires surgical repair (medial collateral ligament [MCL], posterior cruciate ligament[PCL]), chondral defects >2cm, fracture, bilateral knee injury
* Medial conditions that are contraindications to electrical stimulation: Cardiac Pacemaker and Pregnancy
* Participants who are unable to understand procedures of experiment or provide consent (assent/parental permission)

Ages: 14 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 39 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Quadriceps Rate of Torque Development (RTD) Maximum | Change from Baseline Quadriceps RTD at 3 weeks
  slope of the torque-time tracing (change in torque/change in time) (Nm/kg*s-1)
Knee Joint biomechanics during gait (nonlinear) | Change from Baseline nonlinear knee joint biomechanics at 3 weeks
  Sagittal plane (knee flexion) movement variability (calculated using Lyapunov Exponent and approximate entropy)

SECONDARY OUTCOMES:
Quadriceps percent activation | Change from Baseline Quadriceps percent activation at 3 weeks
  Supramaximal electrical stimulus (interpolated twitch technique) used to augment a voluntary muscle contraction
Knee Joint biomechanics during gait (traditional) | Change from Baseline knee joint biomechanics at 3 weeks
  peak external knee flexion moment (Nm/kgm)
Patient reported function | Change from Baseline IKDC at 3 weeks
  International Knee Documentation Committee (IKDC) subjective form
Jumping performance | Change from Baseline single leg hop for distance at 3 weeks
  single leg hop for distance (cm)

CONTACTS AND LOCATIONS:
Overall Officials: Terry L Grindstaff, PhD, PT, ATC, Principal Investigator — Creighton University
Locations (1):
- Creighton University, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No